CLINICAL TRIAL: NCT06710704
Title: A Comparative Study Between Transcutaneous Pulsed Radiofrequency and Corticosteroids Injections in Management of Pain in Lateral Epicondylitis
Brief Title: Transcutaneous Pulsed Radiofrequency and Corticosteroids Injections in Management of Pain in Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Magdy Ahmed Elgazzar, Resident of Anesthesiology,Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264MS267/7/23
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Transcutaneous; Pulsed Radiofrequency; Corticosteroids Injections; Pain; Lateral Epicondylitis
MeSH Terms: conditions — Pain; Tennis Elbow | interventions — Methylprednisolone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous pulsed radiofrequency group (Experimental): Patients underwent transcutaneous pulsed radiofrequency at the affected elbow.
  Interventions: Device: Transcutaneous pulsed radiofrequency
- Control group (Active Comparator): Patients received intraarticular injections of methylprednisolone (40 mg/ml) with 1 ml mepacaine at the point with utmost tenderness in the lateral epicondyle area under aseptic conditions.
  Interventions: Drug: Methylprednisolone and mepacaine

INTERVENTIONS:
Device: Transcutaneous pulsed radiofrequency — Patients underwent transcutaneous PRF at the affected elbow.
  Arms: Transcutaneous pulsed radiofrequency group
Drug: Methylprednisolone and mepacaine — Patients received intraarticular injections of methylprednisolone (40 mg/ml) with 1 ml mepacaine at the point with utmost tenderness in the lateral epicondyle area under aseptic conditions.
  Arms: Control group

SUMMARY:
The aim of the study is to compare between transcutaneous pulsed radiofrequency and corticosteroids injections in management of pain severity, forearm pain, functional disability and patient capability to operate daily activities in patients with lateral epicondylitis

DETAILED DESCRIPTION:
Lateral epicondylitis (LE), or tennis elbow, is the most common elbow pain condition. Pain in the lateral aspect of the elbow, especially the extensor tendon origin (extensor carpi radialis brevis [ECRB] and extensor digitorum communis [EDC]), is the most consistent symptom. It affects up to 3 % of the population and is usually an overload injury that often follows minor and often unrecognized trauma to the extensor forearm muscles of the forearm.

Transcutaneous pulsed radiofrequency treatment is a noninvasive, needleless, painless, office/outpatient treatment that requires no recovery, sedation, or anesthesia. We were encouraged to research transcutaneous pulsed radiofrequency as a treatment option because of favorable outcomes in previous trials. Therefore, transcutaneous pulsed radiofrequency treatment used successfully in a type of orthopedic surgeries, we designed this trial to examine it in the management of pain in lateral epicondylitis.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18-65 years.
* Both sexes.
* Symptomatic lateral epicondylitis for more than 6 months.

Lateral epicondylitis was diagnosed when pain is elicited by two or more of these diagnostic exams:

1. Palpation of the lateral epicondyle.
2. Resisted wrist extension (Thompson test).
3. Chair test. With the shoulder flexed to 60° and the elbow extended, the patient attempts to lift a chair weighing 3.5 kg.

Exclusion Criteria:

* Severe systemic diseases (diabetes or rheumatoid arthritis).
* Cervical radiculopathy.
* Major trauma or prior surgery in the tendon of the elbow.
* Morbid obese patients (body mass index (BMI) of >35 kg/m2).
* Infection at site of injection.
* Bleeding diathesis and coagulopathy.
* Patients who didn't consent to completing visual analog scale , rated tennis elbow evaluation (PRTEE), disabilities of the Arm, Shoulder, and Hand (Quick DASH) questionnaire. and refuse to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Degree of pain. | 12 weeks after treatment
  Assessment of pain severity by visual analog scale (VAS) before treatment and at 2, 4, 8, and 12 weeks after treatment.
  The visual analog scale (VAS) score it has 10-cm scale that represents a continuum between "0 = no pain" and "10 = worst pain."

SECONDARY OUTCOMES:
Forearm pain | 12 weeks after treatment
  Forearm pain wasassessed by patient-rated tennis elbow evaluation (PRTEE).
  The Rated Tennis Elbow Evaluation (PRTEE) was also used to rate the levels of tennis elbow pain and disability from 0 to 10, and consists of 2 subscales:
  Pain subscale - 5 items (0 = no pain, 10 = worst imaginable). Function subscale (0 = no difficulty, 10 = unable to do) Specific activities - 6 items.
Functional disability | 12 weeks after treatment
  Functional disability was assessed by patient-rated tennis elbow evaluation (PRTEE) before treatment and at 2, 4, 8, and 12 weeks after treatment..
  The Rated Tennis Elbow Evaluation (PRTEE) was also used to rate the levels of tennis elbow pain and disability from 0 to 10, and consists of 2 subscales:
  Pain subscale - 5 items (0 = no pain, 10 = worst imaginable). Function subscale (0 = no difficulty, 10 = unable to do) Specific activities - 6 items.
Patient capability | 12 weeks after treatment
  Patient capability to operate daily activities was evaluated using Disabilities of the Arm, Shoulder, and Hand (Quick DASH) questionnaire before treatment and at 2, 4, 8, and 12 weeks after treatment.
  The Quick DASH is a shortened edition of the original DASH result amount. Quick DASH was used to measure of self-rated upper-extremity disability and symptoms before. It is a 11-item and self-report questionnaire that looks at the ability of a patient to perform certain upper extremity activities, patients can rate difficulty and interference with daily life on a 5-point Likert scale (1 being no difficulty, 5 being unable).

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, ElGharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data was available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data was available upon a reasonable request from the corresponding author.